CLINICAL TRIAL: NCT03207802
Title: Necklace-Shaped Sensor for Non-Invasive Measurement of Vital Signs, Thoracic Impedance, ECG, Skin Temperature and Motion
Brief Title: Remotely Monitoring Patients With Chronic Conditions in Their Home
Status: Completed | Type: Observational
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PERM-IRB-001-OCS
Record Dates: First submitted 2017-06-30; First posted 2017-07-05 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2018-01

CONDITIONS: CHF

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Cohort 3: This cohort is living at home with a chronic condition.
  Interventions: Device: Discontinuation of using device

INTERVENTIONS:
Device: Discontinuation of using device — Subject will be instructed to discontinuation of use of device

SUMMARY:
Study will collect data from the home using the CoVa Monitoring System. Data will be captured and retrospectively analysis to determine if the data provided can alert clinician about a patient's declining health.

DETAILED DESCRIPTION:
Study will collect data from the home using the CoVa Monitoring System. Data will be captured and retrospectively analysis to determine if the data provided can alert clinician about a patient's declining health. Data from the CoVa Monitoring System will be compared against electronic health records to determine if the data captured will provide insight into a patient's overall health. Additionally, user compliance will be monitored

ELIGIBILITY:
Inclusion Criteria:

* Chronic Disease including CHF
* Currently receiving home health care
* Recent discharge for a CHF event

Exclusion Criteria:

* Skin reaction to electrodes
* Inability to take measurements due to low BMI

Ages: 22 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving home health care with one or more chronic diseases including CHF
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2017-12-17 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Data correlation | 2-6 months
  Correlation between data collection and potential heart failure event

CONTACTS AND LOCATIONS:
Locations (1):
- Elite Home Health, Texarkana, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No